CLINICAL TRIAL: NCT02358148
Title: Validation of the Simple Acute Coronary Syndrome (SACS) Score and Head-to-Head Comparison of the SACS vs. Modified TIMI vs. HEART ACS Scores
Brief Title: Validation of Simple Acute Coronary Syndrome (SACS) Score
Acronym: SACS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bayfront Health St Petersburg (Other)
Collaborators: Bayfront Health Dade City (Unknown); Community Health Systems (CHS) (Unknown)
Responsible Party: Principal Investigator, Wayne Ruppert, Cardiac Data Specialist and Cardiovascular Clinical Coordinator, Bayfront Health St Petersburg
Other Study IDs: 521-0
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Angina; Myocardial Infarction
Keywords: Acute Coronary Syndrome; Chest Pain; ACS; Risk Stratification Score; HEART Score; Modified TIMI; Coronary Artery Disease; Risk Factors; Myocardial Infarction
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Angina Pectoris; Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- STEMI / NSTEMI: All patients (100%) admitted to the participating hospitals during the study period with the diagnosis of Acute ST Segment Myocardial Infarction (STEMI) or Non-ST Segment Myocardial Infarction (NSTEMI) will be selected for inclusion in the study. In order to assure rapid door-to-reperfusion times, Study Investigators will obtain consent and interview these patients AFTER cardiac catheterization and intervention. A minimum number of 25 STEMI and 25 NSTEMI patients will be enrolled in the study.
- Elective / Non-emergent Cardiac Cath: This group will include both admitted and outpatients, with possible diagnoses of Unstable Angina (UA), Low Risk Chest Pain (LRCP), and those having cardiac catheterization for any other reason (eg: elective, medical clearance for surgery, failed stress test, etc.). To maintain integrity of the study, these patients will be randomly selected, with written consent obtained, prior to cardiac catheterization.

SUMMARY:
This prospective observational study will evaluate and compare the sensitivity and specificity of the Modified TIMI, HEART and SACS Scores for accurately predicting the presence and absence of obstructive coronary artery disease (OCAD) as diagnosed during coronary angiography in the cardiac catheterization suite. In addition, we plan to determine if a variant of SACS, HEART, TIMI, or a hybrid score resulting from combining formulas from two or all three scores yields a new tool that exceeds the predictive performance of all three current models for determining the absence or presence of OCAD.

DETAILED DESCRIPTION:
HISTORY: The Simple Acute Coronary Syndrome (SACS) Score was developed in 2009 by Cardiac Catheterization staff after noting what appeared to be an unacceptable volume of patients presenting with low Modified TIMI Scores (0-2) who were found to have severe Obstructive Coronary Artery Disease (OCAD). The SACS Scoring formula was derived by observing correlations in an estimated 12,000 cases between patients' SYMPTOMS, ECG FINDINGS, CAD RISK FACTOR PROFILES, TROPONIN VALUES and the degree of OCAD discovered during coronary angiography.

The primary objective of the SACS Score is to identify patients who are at high risk for OCAD, with the intent that they will receive diagnostic and interventional measures prior to the occurence of Acute Myocardial Infarction (AMI) or other Major Adverse Coronary Event (MACE).

In a small pilot study conducted in 2009 at St Joseph's Hospital in Tampa, Florida, the SACS Score demonstrated a trend of reliability superior to the Modified TIMI Score for accurately predicting the absence or presence of OCAD. Because the sample size was deemed to be not statistically significant (n=42), the study team concluded that the "SACS Score demonstrates a promising trend, but additional data needs to be collected and analyzed before any definitive conclusions can be drawn."

Since the advent of the St Joseph's study, another ACS / MACE predictive tool, the HEART Score, was introduced by Backus and Six et al of the Netherlands. The HEART Score has been scientifically validated by several studies with results published most recently in the International Journal of Cardiology (2013). Furthermore the studies demonstrated that HEART is superior to the Modified TIMI and GRACE Scores for accurately predicting the probability of MACE.

It is interesting to note that the HEART Score closely resembles SACS, with differences in the scoring formula for ECG findings and the patient's age. Our hypothesis is both scores will demonstrate superior predictability of OCAD, but a hybrid combination of the HEART and SACS formulas may produce a scoring tool that will exceed all three in sensitivity and specificity for predicting the presence or absence of OCAD.

STUDY END POINT for all patients is CARDIAC CATHETERIZATION: The findings obtained during CORONARY ANGIOGRAPHY, and the need for immediate intervention, as dictated by the Interventional Cardiologist.

DATA TO BE COLLECTED: Patient symptoms, history, CAD risk factor profile, 12 Lead ECG findings, Lab results (Troponin, electrolytes, BUN/Creatinine, BNP), and all other data fields necessary to calculate a complete Modified TIMI, HEART and SACS score, Cardiac Cath Lab findings (description of coronary angiography for each vessel) and any Coronary Artery Interventions performed or recommended (PCI, CABG). . A STANDARDIZED DATA COLLECTION FORM has been developed and will be utilized for all patients.

REGRESSION ANALYSIS will result from 126 data points collected from each patient encounter. Relationships between score values and the degree of obstructive CAD present will be established, along with p values and sensitivity / specificity for each scoring system. Recommendations for modifications to currently existing scores, and/or proposals for development of a hybrid scoring system will result from the analysis of this data.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting to the Cardiac Catheterization Lab during the study period.

Exclusion Criteria:

* Patients who refuse / wish to not be included in the study,
* Patients with Wolff-Parkinson-White syndrome with visible Delta waves on the ECG.
* Patients with Renal Failure and abnormally elevated Creatinine >2.0
* Patients with Potassium values >6.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients selected in this study will be patients who are having URGENT (Group 1) or NON-URGENT (Group 2) cardiac catheterization performed:
  Group 1: All (100%) of STEMI / Non-STEMI patients presenting for cardiac catheterization during the study period, with a minumum number of 25 STEMI and 25 NSTEMI patients to be included.
  Group 2: Non-urgent cardiac catheterization patients will be randomly selected, with consents obtained, PRIOR TO elective cardiac catheterization.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Angiographic Findings of Cardiac Catheterization | 30 days from enrollment
  Interventional Cardiologist's Diagnosis resulting from coronary angiography during Cardiac Catheterization - will determine which one of the following SECONDARY OUTCOME categories the patient is placed in:

SECONDARY OUTCOMES:
No CAD noted - no coronary interventions indicated | 30 days from study enrollment
  Diagnostic coronary angiography reveals patient has no discernable coronary artery disease, no coronary artery interventions are indicated.
Mild-moderate CAD noted - no coronary artery interventions are indicated | 30 days from study enrollment
  Diagnostic coronary angiography revealed one or more mild-moderate NON-Obstructive Lesion(s), no invasive intervention (PCI or CABG) indicated at current time.
Obstructive CAD present, no myocardial injury, immediate intervention is indicated | 30 days from study enrollment
  Coronary angiography revealed significant Obstructive Lesion(s) present in one or more coronary artery. TIMI Grade III bloodflow is present, intervention (PCI or CABG revascularization) is indicated now.
Obstructive CAD present with myocardial infarction/ injury | 30 days from study enrollment
  Coronary angiography revealed sub-total or total occlusion with <TIMI Grade III flow in one or more coronary artery, myocardial injury/infarction present, immediate intervention (PCI or CABG) indicated.
No Obstructive CAD present but myocardial damage is evident | 30 days from study enrollment
  Coronary angiography reveals no obstructive CAD is present, but patient has sustained myocardial injury with decreased EF, consistent with vascular event such as vasospasm, Apical Balloon (Tako-Tsubo) Syndrome, Cocaine/Drug induced, or other myocardial injury.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Ruppert, CVT, CCCC, Principal Investigator — Bayfront Health Dade City; Ravi Korabathina, MD, FSCAI, Principal Investigator — Bayfront Health St Petersburg
Locations (2):
- United States (2):
  - Bayfront Health Dade City, Dade City, Florida
  - Bayfront Health St Petersburg, St. Petersburg, Florida

REFERENCES:
- [Result] Macdonald SP, Nagree Y, Fatovich DM, Brown SG. Modified TIMI risk score cannot be used to identify low-risk chest pain in the emergency department: a multicentre validation study. Emerg Med J. 2014 Apr;31(4):281-5. doi: 10.1136/emermed-2012-201323. Epub 2013 Apr 10. PMID 23576231
- [Result] Backus BE, Six AJ, Kelder JC, Bosschaert MA, Mast EG, Mosterd A, Veldkamp RF, Wardeh AJ, Tio R, Braam R, Monnink SH, van Tooren R, Mast TP, van den Akker F, Cramer MJ, Poldervaart JM, Hoes AW, Doevendans PA. A prospective validation of the HEART score for chest pain patients at the emergency department. Int J Cardiol. 2013 Oct 3;168(3):2153-8. doi: 10.1016/j.ijcard.2013.01.255. Epub 2013 Mar 7. PMID 23465250
- See also: Heart Score Netherlands - website — http://heartscore.nl/score